CLINICAL TRIAL: NCT05331547
Title: A Pilot Study Registry of the BioFreedom™ BA9™ Ultra Drug-Coated Coronary Stent for Patients With ST Elevation Myocardial Infarct (STEMI) Undergoing Percutaneous Coronary Intervention (PCI)
Brief Title: BioFreedom™ BA9™ Ultra
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Biosensors International (Other)
Responsible Party: Sponsor
Other Study IDs: UW 21-385
Record Dates: First submitted 2021-08-19; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Death; Myocardial Infarction; Revascularization
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- BioFreedom BA9 (SS) Ultra DCS: STEMI patients treated with one or several BioFreedom stent(s)
  Interventions: Device: BioFreedom BA9 (SS) Ultra DCS

INTERVENTIONS:
Device: BioFreedom BA9 (SS) Ultra DCS — BioFreedom Ultra stent for treatment of STEMI patients. Besides, in patients who are clinically indicated for a stage procedure, we aim to assess the angiographic and endovascular healing of BioFreedom Ultra stent at one month
  Other Names: optic coherence tomography (OCT)

SUMMARY:
The purpose of the study is to assess the safety and efficacy of the BioFreedom Ultra stent for treatment of STEMI patients. Besides, in patients who are clinically indicated for a stage procedure, Investigators aim to assess the angiographic and endovascular healing of BioFreedom Ultra stent at one month

This is a prospective, single center, post marketing registry. Investigators aim to recruit 50 patients. All enrolled patients will be followed up for 12 months.

Restudy Subgroup For subjects who are clinically indicated for staged procedure, they will be recruited into restudy subgroup. Restudy angiogram of target lesion will be performed at 28 (±7) days. Intravascular OCT will be performed.

The primary endpoint is target lesion failure (TLF) defined as composite of cardiovascular death, target-vessel related myocardial infarction (Q-wave and non-Q-wave), or ischemia-driven target lesion revascularization within 12 months (device-oriented outcome per ARC definitions)

The co-primary endpoint in subjects who require stage procedure is stent strut coverage (degree of endothelialisation) as assessed by optic coherence tomography (OCT) at one month

Secondary endpoints include

1. All-cause mortality
2. Cardiovascular death (cardiovascular and undetermined)
3. The composite of cardiovascular death, Target Lesion (TL)-related myocardial infarction and TL-related definite or probable stent thrombosis at one year.
4. Stroke disabling and non-disabling ARC definition
5. Myocardial infarction
6. ARC Stent thrombosis
7. Clinically driven TLR at any follow-up time point
8. Clinically driven target vessel revascularization
9. Any revascularization within 12 months following the index procedure, unless they are planned within the 1st month
10. Bleeding per BARC criteria

    For subjects in restudy subgroup
11. Restudy angiographic result (QCA)
12. OCT parameters including neointimal volume, neointimal area etc

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death and disability worldwide. One severe manifestation of CAD is acute ST elevation myocardial infarction (STEMI) which is commonly due to atherothrombosis of major epicardial coronary artery. The treatment aim of STEMI is emergent reperfusion of blocked coronary artery by mechanical or pharmacological means. Percutaneous coronary intervention (PCI) with stent implantation of obstructive coronary lesions has been shown to improve patients' survival and outcome.

Early generation drug-eluting stents (DES), namely, sirolimus-eluting stents and paclitaxel-eluting stents, have been compared with bare-metal stents (BMS) in the clinical setting of STEMI in several randomized controlled trials and consistently showed a reduction in major adverse cardiac events (MACE) mainly related to a lower risk of repeat revascularization procedures [1-6]. However, vessel healing is delayed with evidence of chronic inflammation related at least in part to the persistence of durable polymer components in patients with acute STEMI [7] after implantation of a DES compared to a BMS DES as opposed to BMS implanted into a pro-thrombotic, inflammatory milieu of ruptured plaques in STEMI patients may lead to aneurysmal changes of the adjacent vessel wall. Moreover, DES implanted into STEMI lesions have been associated with a higher frequency of incompletely apposed struts and uncovered struts as assessed by OCT compared with DES implanted into stable lesions [7]. These data suggest a significantly increased risk of late thrombotic complications related to DES. In recent years, newer-generation devices with drug release from durable or biodegradable polymer surface coating may provide the basis for improved biocompatibility and vascular healing [8]. The EXAMINATION (clinical Evaluation of the Xience-V stent in Acute Myocardial INfArcTION) and COMFORTABLE-AMI (Comparison of Biolimus Eluted From an Erodible Stent Coating With Bare Metal Stents in Acute ST-Elevation Myocardial Infarction) trials have tested the efficacy of everolimus eluted from durable polymer (everolimus-eluting stent [EES]) and of biolimus A9 eluted from biodegradable polymer (biolimusA8-eluting stent [BES]) stents versus BMS, respectively, in an all-comer STEMI population [9-12]. Whereas the EXAMINATION trial showed a significant reduction in stent thrombosis with the EES (0.9% vs. 2.5%, p = 0.019), the COMFORTABLE-AMI trial demonstrated a significant reduction in MACE with the BES (4.3% vs. 8.7%, p = 0.004) compared with BMS at 1 year [12].

In view of concerns over long term safety of DES polymer, third generation of stents that still release drug but without polymer are being developed. The BioFreedom DCS Coronary Stent Delivery System is comprised of three key components including 1) a 316 L stainless steel bare metal stent platform which has been modified with a proprietary surface treatment resulting in a selectively micro-structured, abluminal surface. The selectively micro-structured surface allows 2) Biolimus A9 (drug) adhesion to the abluminal surface of the stent without the use of a polymer or binder.

The BioFreedom First In Man (FIM) trial was a prospective, single blinded, randomized clinical trial to evaluate the safety and effectiveness of a low and standard dose BioFreedom Biolimus A9 Drug-Eluting Coronary Stent Delivery System compared with a Taxus® Liberté® control arm for the treatment of stenotic lesions in native coronary arteries [13]. The BioFreedom FIM trial documented, that the BioFreedom (BFD) stent was non-inferior to the CE-mark approved Taxus Liberté Paclitaxel Eluting stent (PES) for the angiographic endpoint "in-stent late lumen loss" at 12 months (BFD 0.17mm vs. PES 0.35mm; p=0.001 for non-inferiority; p=0.11 for superiority). Despite a numerically better late lumen loss for the BFD, superiority was not reached. Both stents showed similar clinical outcomes at 12 months with MACE rates of 6.1% (BFD) vs. 5.5% (PES) (p=0.98), and of 23.8% (BFD) vs. 20.3% (PES) at 5 years (p=0.67). No ARC definite/probable stent thrombosis occurred in either arm. These results demonstrated that the BFD stent has comparable angiographic efficacy at 1 year and similar long-term safety outcomes as the PES out to 5 years.

Later on, The LEADERS FREE trial [14] was a prospective, randomized, double-blind trial to evaluate the safety and efficacy of the BioFreedom polymer-free and carrier-free drug-coated stent compared with a bare-metal stent (BMS) in patients with increased bleeding risk. 2,466 patients were enrolled at 68 sites in 20 countries from December 2012 through May 2014, with 1,239 randomly assigned to the BioFreedom stent, and 1,227 randomly assigned to the bare-metal stent. All patients were prescribed one month of dual antiplatelet therapy. Inclusion criteria were designed to create a patient population with high bleeding risk (or otherwise considered as candidates for a BMS as opposed to a DES, and not considered suitable for prolonged dual antiplatelet therapy). Patients with coronary artery disease and a clinical indication for PCI were eligible if they met one or more inclusion criteria. The trial was powered to determine whether the BioFreedom stent was non-inferior to the bare-metal stent in 2-years outcomes according to the primary safety endpoint. If non-inferiority was shown, the safety endpoint would then be tested for superiority. The primary safety endpoint was a composite of cardiac death, MI, and definite or probable stent thrombosis at two different time point: a 390 and a 790-days time point. The primary efficacy endpoint was incidence of clinically-driven target-vessel revascularization (CI-TLR) at 390 and 790 days. 2,432 patients underwent PCI, and 2,386 (98.1%) were followed until death or 730 days, with follow-up visits at 30 days and 1 year, and either on-site or telephone follow-up at 2 months, 4 months, and 2 years.

The primary safety endpoint (cumulative incidence of cardiac death, MI, or stent thrombosis through 390 days) occurred in 112 patients (9.4%) in the BioFreedom group and 154 patients (12.9%) in the BMS group (P < 0.001 for non-inferiority and P = 0.005 for superiority). The significantly lower incidence of the composite safety endpoint in the BioFreedom group was due largely to a lower rate of MI, with 72 patients (6.1%) vs. 104 patients (9.0%) experiencing any MI (P = .01).

In the BioFreedom group, 50 patients (4.2%) died from cardiac causes compared with 63 cardiac deaths (5.3%) in the BMS group. Rates of stent thrombosis were similar in the two groups, with 24 patients (2.0%) vs. 26 patients (2.2%) experiencing thrombosis through 390 days.

The primary efficacy endpoint (CI-TLR through 390 days) occurred in 59 patients (5.1%) in the BioFreedom group and 113 patients (9.8%) in the BMS group (P <.001). Bleeding was high in both groups, as expected, with 215 BioFreedom patients (18.1%) vs. 225 BMS patients (19.1%) experiencing bleeding at 1 year.

On the whole, BioFreedom stent was superior to a bare metal stent both in efficacy and safety, when used with a 1-month regimen of dual antiplatelet therapy in patients with high bleeding risk following PCI. Biofreedom stent is currently CE Mark approved to be used in CAD. It is commercially available in public and private hospitals in Hong Kong.

The Biofreedom Ultra stent is the latest version of Biofreedom stent with improved stent design. Contrary to Biofreedom DCS, the Biofreedom Ultra is made of Cobalt chromium which is a more commonly used material in DES nowadays. Therefore, Biofreedom ultra has better strength and can be manufactured to have thinner struts which enhanced its flexibility and crossibility. The Leaders Free III trial is a single arm trial involving 400 patients with high bleeding risk. Patients were implanted Biofreedom ultra stents and all were given one month dual antiplatelet therapy (DAPT). Compared with previous data, Biofreedom ultra is non-inferior to Biofreedom DCS and is superior to BMS in efficacy and safety. Currently, Biofreedom ultra has obtained CE Mark for use in CAD. It is also approved for commercial use in hospitals in Hong Kong.

Objective and purpose

The purpose of the study is to assess the safety and efficacy of the BioFreedom Ultra stent for treatment of STEMI patients. Besides, in patients who are clinically indicated for a stage procedure, investigators aim to assess the angiographic and endovascular healing of BioFreedom Ultra stent at one month

Trial Design

This is a prospective, single center, post marketing registry. Investigators aim to recruit 50 patients. All enrolled patients will be followed up for 12 months.

Restudy Subgroup For subjects who are clinically indicated for staged procedure, they will be recruited into restudy subgroup. Restudy angiogram of target lesion will be performed at 28 (±7) days. Intravascular OCT will be performed.

The primary endpoint is target lesion failure (TLF) defined as composite of cardiovascular death, target-vessel related myocardial infarction (Q-wave and non-Q-wave), or ischemia-driven target lesion revascularization within 12 months (device-oriented outcome per ARC definitions)

The co-primary endpoint in subjects who require stage procedure is stent strut coverage (degree of endothelialisation) as assessed by optic coherence tomography (OCT) at one month

Secondary endpoints include

1. All-cause mortality
2. Cardiovascular death (cardiovascular and undetermined)
3. The composite of cardiovascular death, Target Lesion (TL)-related myocardial infarction and TL-related definite or probable stent thrombosis at one year.
4. Stroke disabling and non-disabling ARC definition
5. Myocardial infarction
6. ARC Stent thrombosis
7. Clinically driven TLR at any follow-up time point
8. Clinically driven target vessel revascularization
9. Any revascularization within 12 months following the index procedure, unless they are planned within the 1st month
10. Bleeding per BARC criteria

    For subjects in restudy subgroup
11. Restudy angiographic result (QCA)
12. OCT parameters including neointimal volume, neointimal area etc

Selection and Withdrawal of Subjects

The registry is open to all consecutive patients (male or female) presenting with STEMI and treated with one or more BioFreedom BA9 (SS) Ultra DCS.

Patients will be asked to give consent after the index procedure

Each patient is free to withdraw from the registry at any time and without reason, and without influence on their further medical treatment or relationship to their physicians. Once the patient is withdrawn, they will be followed per institutional standard of care.

Every effort will be made by the investigator to keep the patient in the registry; however, should the patient decide to withdraw, the investigator is responsible for reporting the observations thoroughly, and completing the final evaluations and eCRFs. The primary reason for the early withdrawal must be documented on the Study Exit case report form.

For patients who withdraw their consent after the commencement of any PCI procedure, a final follow-up either by phone or clinic visit will be conducted.

Treatment of Subjects, study procedures and follow up

ST-elevation Myocardial Infarction (STEMI) patients who have received BioFreedomBA9 (SS) Ultra DCS stents and who meet the eligibility criteria will be invited to join the registry and asked to sign a consent form prior to inclusion into the study. The details will be explained by the cardiologist with the patient information sheet. Eligible patients who sign the consent form which includes a data release section, will be enrolled into the registry.

A copy of the signed consent form will be given to the patient and a copy will be filed in their medical file.

The patient can be enrolled after they have received the BioFreedom BA9 (SS) DCS stent and have fully signed the consent and data release form. Enrollment is completed when they are also assigned a patient ID. Upon patient enrolment, the relevant patient data will be entered in the case report form (CRF). These data are routinely collected in normal clinical practice and include:

1. Confirmation of signing the consent form
2. Relevant medical history
3. Medication
4. PCI indications
5. Eligibility
6. Notes on the PCI procedure, number of stents implanted, BioFreedom BA9 (SS) Ultra DCS stent details and any procedural complications will be entered in the CRF.
7. Restudy angiographic and intravascular imaging result (For restudy subgroup only)

Patients will be followed after hospital discharge up to 12 months after the index procedure.

These follow-ups consist of telephone contacts or clinic visits, if part of routine hospital practice, to obtain information regarding medication use, hospitalizations, TLFs, all cardiac and procedure related events and serious adverse events at 1,4, and 12 months.

1. Follow up 30 days Post-Procedure (± 7 days) - Telephone An assessment of medication intake and any adverse event will be obtained via telephone contact. Information will be requested from the patient regarding their medication intake inclusive of antiplatelet therapy treatment prescribed by the physician: start and stop date, reason for discontinuation, duration and type of therapy prescribed.
2. Follow up 4 months (± 10 days) Post-Procedure - Telephone An assessment of medication intake and any adverse event will be obtained via telephone contact. Information will be requested from the patient regarding their medication intake inclusive of antiplatelet therapy treatment prescribed by the physician: start and stop date, reason for discontinuation, duration and type of therapy prescribed.

3 Follow up 12 months (± 10 days) Post-Procedure - Telephone or On-Site Visit An assessment of medication intake and any adverse event will be obtained via telephone contact or on-site visit. Information will be requested from the patient regarding their medication intake inclusive of antiplatelet therapy treatment prescribed by the physician: start and stop date, reason for discontinuation, duration and type of therapy prescribed.

Assessment of Efficacy

N/A

Assessment of Safety

Safety of the patients participating in this registry will be monitored throughout the study using the Adverse Event reporting process to identify real and potential safety issues.

An adverse event is any untoward medical occurrence, unintended disease or injury or untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device.

An adverse event (AE) is serious if the event led to death or led to serious deterioration in the health of a patient resulting in a life-threatening illness or injury, a permanent impairment of a body structure or a body function, in patients' hospitalization or prolongation of existing hospitalization and/or in medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function.

Any serious adverse event (SAE) experienced by the enrolled patients will be collected throughout the registry duration

Statistics

Descriptive analysis of baseline and 12-month data will be calculated. Continuous data of demographic and clinical characteristics are expressed as numbers with mean and standard deviation, whereas categorical data are expressed as counts and percentages. Differences in the distributions of continuous variables will be examined using t tests as appropriate. The categorical variables will be analysed using the χ2 or Fisher test.

The number and percentage of clinical endpoints will be described. All clinical endpoints during the course of the study will be adjudicated and analysed.

All the tests are 2-sided with 95% confidence interval and statistical significance is accepted at the P<0.05 level. All analyses will be performed using IBM SPSS Statistics Version 23.

This is an investigator-initiated study. OCT Core Lab, monitoring costs will be supported by unrestricted grant from Biosensors International. No other sponsorship or funding exists.

ELIGIBILITY:
Inclusion Criteria:

1. STEMI patients treated with one or several BioFreedom stent(s)
2. Patients who agree to comply with the follow up requirements.
3. Patients with a life expectancy of > 1 year at time of consent.
4. Patients eligible to receive dual anti platelet therapy (DAPT). The establishment of the DAPT regimen is at the physician's discretion.

Exclusion Criteria:

1. Patients in cardiogenic shock
2. Any out of hospital cardiac arrest
3. Glasgow score < 15
4. Patients unable or unwilling to give documented informed consent
5. Patients taking part in another interventional trial which has not completed follow-up for the primary endpoint
6. Pregnant or breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A prospective, single center, post marketing registry. We aim to recruit 50 patients. All enrolled patients will be followed up for 12 months.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-07-21 (Estimated); Study Completion 2024-01-21 (Estimated)

PRIMARY OUTCOMES:
Stent strut coverage (degree of endothelialisation) | At one month
  Require stage procedure as assessed by optic coherence tomography (OCT) at one month
Target lesion failure (TLF) | Within 12 months (device-oriented outcome per ARC definitions)
  Target-vessel related myocardial infarction (Q-wave and non-Q-wave), or ischemia-driven target lesion revascularization

SECONDARY OUTCOMES:
BioFreedom Ultra stent at one month | At one month
  For subjects in restudy subgroup
  1. Restudy angiographic result (QCA)
  2. OCT parameters including vessel length density: (mm-1), perfusion density: (white pixels/(white + black pixels)] × 100
MACE | Within 12 months
  Secondary endpoints include
  1. All-cause mortality (number in P value)
  2. Cardiovascular death (cardiovascular and undetermined) (number in P value)
  3. The composite of cardiovascular death, Target Lesion (TL)-related myocardial infarction and TL-related definite or probable stent thrombosis at one year. (number in P value)
  4. Stroke disabling and non-disabling ARC definition (number in P value)
  5. Myocardial infarction (number in P value)
  6. ARC Stent thrombosis (number in P value)
  7. Clinically driven TLR at any follow-up time point (number in P value)
  8. Clinically driven target vessel revascularization (number in P value)
  9. Any revascularization within 12 months following the index procedure, unless they are planned within the 1st month (number in P value)
  10. Bleeding per BARC criteria (number in P value)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No